CLINICAL TRIAL: NCT05958589
Title: Efficacy and Safety of General Anesthesia With Caudal Block for Inguinal Hernioplasty in Children: a Randomized Controlled Trial
Brief Title: Caudal Block for Inguinal Hernioplasty in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Mihaela Preveden, Research Assistant, University of Novi Sad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05689/25-2
Record Dates: First submitted 2023-07-07; First posted 2023-07-24 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain
Keywords: general anesthesia; caudal block; pain; hemodynamic parameters
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Levobupivacaine; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia + caudal block (Experimental): General anesthesia with intravenous anesthetic propofol (2-3 mg/kg), opioid analgesic fentanyl (1-1.5 mcg/kg), and muscle relaxant rocuronium - bromide (0.6-1 mg/kg), in combination with a single shot caudal block with levobupivacaine 0.25% (2.5 mg/kg; maximal dose 75 mg).
  Interventions: Drug: Caudal block with levobupivacaine; Drug: General anesthesia; Procedure: Inguinal hernioplasty
- General anesthesia (Active Comparator): General anesthesia with intravenous anesthetic propofol (2-3 mg/kg), opioid analgesic fentanyl (1-1.5 mcg/kg), and muscle relaxant rocuronium - bromide (0.6-1 mg/kg)
  Interventions: Drug: General anesthesia; Procedure: Inguinal hernioplasty

INTERVENTIONS:
Drug: Caudal block with levobupivacaine — After the introduction of general anesthesia, a single shot caudal block will be performed with levobupivacaine 0.25% (2.5 mg/kg; maximal dose 75 mg).
  Arms: General anesthesia + caudal block
Drug: General anesthesia — On the day of operation all patients will recieve midazolam 0.5 mg/kg (maximum dose 15 mg) orally. Induction of anesthesia will be the same for all patients and consist of intravenous anesthetic propofol (2-3 mg/kg), opioid analgesic fentanyl (1-1.5 mcg/kg), and muscle relaxant rocuronium - bromide (0.6-1 mg/kg). The airway will be obtained by placing a laryngeal mask (I-gel®).
Procedure: Inguinal hernioplasty — Elective inguinal hernioplasty

SUMMARY:
This is a prospective, randomized, controlled clinical study designed to determine the effectiveness of caudal block combined with general anesthesia in providing intra- and postoperative analgesia, and its effect on hemodynamic stability and drug consumption.

DETAILED DESCRIPTION:
This prospective, randomized, controlled clinical study will include 70 boys aged 3-5 years scheduled for inguinal herniorrhaphy. Participants will be randomized in 1:1 ratio into two groups. The first group will receive general anesthesia for surgery, while the second group will receive general anesthesia in combination with caudal block. Postoperative pain, hemodynamic parameters and total consumption of all medicaments in the perioperative period will be monitored. Complications and side effects of drugs will be observed as well.

ELIGIBILITY:
Inclusion Criteria:

* boys between 3 to 5 years old
* scheduled for elective inguinal hernioplasty
* without comorbidities and chronic therapy, ASA class I
* body mass and growth normal for the given age
* no allergies
* no congenital anomalies and birth complications

Exclusion Criteria:

* emergency surgeries
* surgeries longer than 60 minutes
* acute infections with leucocytosis/leucopenia
* acute or chronic diseases
* deformities and disorders of spine and nervous system
* allergies
* pilonidal cyst and/or inflammation in sacral region

Ages: 3 Years to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 5 hours
  Postoperative pain level measured using the visual analog scale (VAS)
Postoperative pain | 5 hours
  Postoperative pain level measured using the Wong-Baker Faces pain rating scale

SECONDARY OUTCOMES:
Blood pressure | 5 hours
  Noninvasive measurement of systolic and diastolic blood pressure
Heart rate | 5 hours
  Heart rate measured with electrocardiogram

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for health care of children and youth of Vojvodina, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No